CLINICAL TRIAL: NCT04233528
Title: Evaluation of Systemic Microvascular Endothelial Function in Metabolically Healthy Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CAAE 13959019.0.0000.5272
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Dyslipidemias
Keywords: laser speckle contrast imaging
MeSH Terms: conditions — Obesity; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy volunteers (Experimental): metabolically healthy eutrophic individuals (BMI ≥18.5 and <25 kg / m2) without any IDF criteria for metabolic syndrome
  Interventions: Diagnostic Test: Evaluation of systemic skin microvascular endothelial function
- metabolically healthy obesity (Experimental): obese individuals (BMI ≥ 30.0 kg / m2) meeting the criteria for metabolically healthy obesity
  Interventions: Diagnostic Test: Evaluation of systemic skin microvascular endothelial function
- metabolically unhealthy obesity (Experimental): volunteers diagnosed with metabolically unhealthy obesity
  Interventions: Diagnostic Test: Evaluation of systemic skin microvascular endothelial function

INTERVENTIONS:
Diagnostic Test: Evaluation of systemic skin microvascular endothelial function — Laser-based method for evaluating non-invasive, operator-independent systemic microvascular function that detects microvascular flow in the skin for the evaluation of systemic vascular endothelial function.

SUMMARY:
Obesity is known to be a risk factor for cardiovascular disease (CVD), type 2 diabetes mellitus, gastrointestinal tract disease, respiratory problems (such as obstructive sleep apnea), joint and muscle problems, reproductive disorders, depression and cancer.

However, recently a new classification has emerged about obesity, the metabolically healthy obesity (MHO). According to the definition of the term, MHO represents obesity that occurs segregated from the metabolic syndrome criteria defined by the International Diabetes Federation (IDF). However, as there is still disagreement about the definition of MHO, the cardiovascular risk of these individuals is also uncertain. This phenotype may present as an intermediate risk between metabolically healthy normal-weight individuals and metabolically unhealthy obese individuals (MUO) or as a transition stage of the disease; when evolving to MUO, represents a higher risk of developing CVDs.

The hypothesis of the present study is that obese individuals classified as metabolically healthy have worse vascular endothelial function when compared to non-obese individuals, demonstrating increased cardiovascular risk even in this subgroup considered "low risk". The detection of endothelial dysfunction in metabolically healthy obese may help in the prevention, treatment and follow-up of these individuals, aiming to reduce the development and morbidity and mortality of CVD.

In the present study, the investigators will use a laser-based method for evaluating non-invasive, operator-independent systemic microvascular function that detects microvascular flow in the skin for the evaluation of systemic vascular endothelial function.

ELIGIBILITY:
Inclusion Criteria:

• obese individuals (BMI ≥ 30.0 kg / m2) meeting the criteria for metabolically healthy obesity

Exclusion Criteria:

* Pregnancy or lactation.
* Endocrine disorders except diabetes, cardiovascular disease except systemic arterial hypertension, autoimmune diseases, malignant neoplasms.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Baseline and post-iontophoresis of acetylcholine endothelium-dependent skin microvascular reactivity | Microvascular reactivity will be evaluated after a 20-minute rest in the supine position in a temperature-controlled room.
  Evaluation of systemic microvascular reactivity induced by endothelium-dependent agents. Microvascular reactivity will be evaluated using a non-invasive and operator -independent methodology, named laser speckle contrast imaging, coupled with skin iontophoresis of vasodilator agents. Cutaneous microvascular flow will be measured in arbitrary perfusion units, divided by mean arterial pressure, to yield cutaneous vascular conductance.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No